CLINICAL TRIAL: NCT00538174
Title: A Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Dapagliflozin in Diabetic Japanese Subjects
Brief Title: Phase I Multiple-Ascending Dose (Japan)
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-025
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): 2.5 mg
  Interventions: Drug: Dapagliflozin
- Arm 2 (Experimental): 10 mg
  Interventions: Drug: Dapagliflozin
- Arm 3 (Experimental): 20 mg
  Interventions: Drug: Dapagliflozin
- Arm 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, once daily up, to 14 days
  Arms: Arm 1; Arm 2; Arm 3
Drug: placebo — Tablets, Oral, 0 mg, once daily, up to 14 days
  Arms: Arm 4

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) following once daily oral doses of 2.5, 10, and 20 mg of dapagliflozin in diabetic Japanese subjects administered for 14 days

ELIGIBILITY:
Inclusion Criteria:

* Japanese male and female subjects
* Ages 20 to 70 years old
* Established diagnosis of T2DM
* BMI < 32 kg/m2
* Fasting glucose ≤ 240 mg/dL, while on antidiabetic diet alone
* HbA1C 6.0 - 10.0%

Exclusion Criteria:

* Symptomatic T2DM defined as polyuria and/or polydipsia within 2 months of enrollment
* History of diabetic ketoacidosis or hyperosmolar nonketotic syndrome
* History of incontinence or bladder dysfunction including nocturia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
AEs, vital signs & physical exam | scr, Days -3, -1, 1, 2, 7, 12, 13, 14, 15, 21
ECGs | scr, Days -1, 1, 2, 7, 12, 13, 14, 15, 21
Clinical labs | scr, Days -1, 2, 7, 12, 14, 15, 21
Urine safety markers | Days -1, 1, 14

SECONDARY OUTCOMES:
24 hr PK blood & urine samples | Days 1 & 14
Serum glucose, serum insulin, serum c-peptide | Days -1, 1, 14
Serum fructosamine | Days -1, 14, 4 h
OGTT | Days -2, 13 (after 10 h fast)
24h urine | Days -1, 1 & 14 for glucose, creatinine & calcium

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers K.K.
Locations (1):
- Local Institution, Suita, Osaka, Japan

REFERENCES:
- [Result] Kasichayanula S, Chang M, Hasegawa M, Liu X, Yamahira N, LaCreta FP, Imai Y, Boulton DW. Pharmacokinetics and pharmacodynamics of dapagliflozin, a novel selective inhibitor of sodium-glucose co-transporter type 2, in Japanese subjects without and with type 2 diabetes mellitus. Diabetes Obes Metab. 2011 Apr;13(4):357-65. doi: 10.1111/j.1463-1326.2011.01359.x. PMID 21226818